CLINICAL TRIAL: NCT03930836
Title: Implementation of a New Interactive Interface Applying Motor Skill Learning Principles to Generate Motor, Functional and Neuroplastic Changes During High and Low Dosage Interventions in Children With Cerebral Palsy
Brief Title: Implementation of a New Motor Skill Learning Therapeutic Device in Children With Cerebral Palsy Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, Yannick Bleyenheuft, Professor, Université Catholique de Louvain
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B403201316810c
Record Dates: First submitted 2018-06-21; First posted 2019-04-29 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Cerebral Palsy
Keywords: motor function; motor skill learning
MeSH Terms: conditions — Cerebral Palsy | interventions — Occupational Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): high/low dosage intervention, intensive or not (motor function rehabilitation)
  Interventions: Behavioral: Hand Arm Bimanual Intensive Therapy Including Lower Extremities; Behavioral: Conventional physical and occupational therapy
- interface group (Experimental): high/low dosage intensive intervention using the interactive interface (motor function rehabilitation)
  Interventions: Behavioral: Hand Arm Bimanual Intensive Therapy Including Lower Extremities

INTERVENTIONS:
Behavioral: Hand Arm Bimanual Intensive Therapy Including Lower Extremities — Intensive intervention focusing on a constant bimanual coordination with a lower extremities and trunk control stimulation during play and functional activities. 50% of therapeutic time will be performed using the new interactive interface
Behavioral: Conventional physical and occupational therapy — Conventional therapy (physical and occupational therapy) is mainly based on neurodevelopmental therapeutic principles. 50% of therapeutic time will be performed using the new interactive interface
  Arms: control group

SUMMARY:
Study of the efficiency of a new interactive interface to apply all the therapeutic principles of motor skill learning used in high dosage intensive interventions. Investigation of its effects on motor, functional and neuroplastic changes in children after high and low dosage intensive interventions using or not the interface.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of unilateral cerebral palsy
* MACS level I, II or III
* GMFCS level I, II, III

Exclusion Criteria:

* unstable seizure
* cognitive deficit that prevent understanding of simple games
* botulinic toxin injection, surgery, or another unusual intervention in the 6 months preceding the study and for the duration of the study

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 64 (Actual)
Dates: Start 2018-06-14 (Actual); Primary Completion 2020-06-20 (Actual); Study Completion 2020-07-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline Assisting Hand Assessments score at 1 week post-camp | pre-camp (1 week before), post-camp (1 week after), 3 months follow-up
  The Assisting Hand Assessment has been developped to measure and describe the efficacy of use of the affected hand of children with unilateral cerebral palsy bimanual activity performance. This is a standardized criterion-referenced test. It is conducted as a recorded semi-structured play session using specific objects usually used in a bimanual manner. With twenty-two test items, the child's performance is measured and obtain a sum score measure and a scaled score (percent scale).
Change from baseline 6 Minutes Walking Test score at 1 week post-camp | pre-camp (1 week before), post-camp (1 week after), 3 months follow-up
  Measurement developped to assess the exercise tolerance and walking abilities by asking the patient to walk as much as possible during 6 minutes in a 30 meters long corridor

SECONDARY OUTCOMES:
Change from baseline Box and Blocks test score at 1 week post-camp | pre-camp (1 week before), post-camp (1 week after), 3 months follow-up
  Test measuring hand function through the number of blocks transported in 1 minute from one part an other of a box placed in front of the child. Each hand tested separately
Change from baseline Jebsen-Taylor Test of Hand Function score at 1 week post-camp | pre-camp (1 week before), post-camp (1 week after), 3 months follow-up
  Measure of hand function/dexterity, through 7 activities simulating daily life activities. Each hand is tested separately and time to complete each activity is reported using a stopwatch.
Change from baseline Modified Cooper test at 1 week post-camp | pre-camp (1 week before), post-camp (1 week after), 3 months follow-up
  Measurement of the stereognosis abilities.16 objects are placed in the hand and the child has to recognise the object only by touch. both hands are tested separately and time to recognise the objects is reported using a stopwatch
Change from baseline ABILHAND-Kids questionnaire score at 1 week post-camp | pre-camp (1 week before), post-camp (1 week after), 3 months follow-up
  questionnaire measuring performance of the child in daily life activities focusing on the upper extremities.
Change from baseline ACTIVLIM-CP questionnaire score at 1 week post-camp | pre-camp (1 week before), post-camp (1 week after), 3 months follow-up
  questionnaire measuring performance of the child in daily life activities focusing on upper and lower extremities.
Change from baseline ABILOCO-Kids questionnaire at 1 week post-camp | pre-camp (1 week before), post-camp (1 week after), 3 months follow-up
  questionnaire measuring performance of the child in daily life activities focusing on the lower extremities.
Change from baseline Pediatric Evaluation of Disability Inventory score at 1 week post-camp | pre-camp (1 week before), post-camp (1 week after), 3 months follow-up
  questionnaire measuring performance of the child in daily life activities focusing on the upper extremities and lower extremities. Only the self-care domain will be assessed here
Change from baseline Canadian Occupational Performance Measure scores at 1 week post-camp | pre-camp (1 week before), post-camp (1 week after), 3 months follow-up
  The Canadian Occupational Performance Measure is a measure designed to capture the patient's self-perception of performance in everyday living, over time. It consist of a semi-structured interview were the patient elicits daily life activities performed with difficulties (self-care, nutrition, transfer, household management, school, work, transport, leisure, etc). Five activities are then chosen as the most important to improve and score on a 1 to 10 scale based on the actual patient's performance and satisfaction levels.
Change from baseline MHAVIE-child questionnaire score at 1 week post-camp | pre-camp (1 week before), post-camp (1 week after), 3 months follow-up
  Questionnaire measuring social participation

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Neuroscience, Université catholique de Louvain, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Saussez G, Bailly R, Araneda R, Paradis J, Ebner-Karestinos D, Klocker A, Sogbossi ES, Riquelme I, Brochard S, Bleyenheuft Y. Efficacy of integrating a semi-immersive virtual device in the HABIT-ILE intervention for children with unilateral cerebral palsy: a non-inferiority randomized controlled trial. J Neuroeng Rehabil. 2023 Jul 29;20(1):98. doi: 10.1186/s12984-023-01218-4. PMID 37516873